CLINICAL TRIAL: NCT00627042
Title: An Open Label, Multicenter, Phase 2 Study Evaluating the Safety and Efficacy of IMC-1121B as First Line Monotherapy in Patients With Unresectable Hepatocellular Cancer
Brief Title: Study of IMC-1121B (Ramucirumab) in Participants With Liver Cancer Who Have Not Previously Been Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13922; CP12-0710 (Other: ImClone Systems); I4T-IE-JVBQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-02-18; First posted 2008-02-29 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver disease; Neoplasms; Liver neoplasms; Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases; Neoplasms; Liver Neoplasms | interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramucirumab (IMC-1121B) (Experimental)
  Interventions: Biological: Ramucirumab (IMC-1121B)

INTERVENTIONS:
Biological: Ramucirumab (IMC-1121B) — Participants will receive ramucirumab (IMC-1121B) at 8 milligrams per kilogram (mg/kg) administered over 1 hour every other week (every 14 days). Treatment will continue until there is evidence of disease progression, intolerable toxicity, or other withdrawal criteria are met.
  Other Names: Ramucirumab; IMC-1121B; LY3009806

SUMMARY:
A study to determine how long ramucirumab (IMC-1121B) will stop cancer from growing in participants with liver cancer that cannot be treated with surgery.

DETAILED DESCRIPTION:
Inhibition of angiogenesis is considered a promising approach to the treatment of cancer. Members of the vascular endothelial growth factor (VEGF) family and the VEGF receptor-2 (VEGFR-2) are important mediators of angiogenesis and are likely important therapeutic targets in advanced hepatocellular cancer (HCC).

Angiogenesis appears integral to HCC development and pathogenesis. Angiogenesis inhibition has been efficacious in both in vitro and in vivo HCC models and results of clinical studies also suggest potential to inhibit disease growth.

Ramucirumab is a fully human monoclonal antibody (MAb) that specifically binds to the extracellular domain of VEGFR-2 with high affinity. Phase 1 studies currently nearing completion have demonstrated safety and tolerability at clinically relevant doses, with preliminary evidence of clinical efficacy in a variety of human cancers.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have histologically-confirmed, unresectable HCC
* The participant has at least one unidimensionally-measurable target lesion [≥ 2 centimeters (cm) with conventional techniques, or ≥ 1 cm by spiral computed tomography (CT) or magnetic resonance imaging (MRI)], as defined by Response Evaluation Criteria in Solid Tumors (RECIST). Target lesion(s) must not lay within a previously irradiated, ablated, or chemoembolized area. If a target lesion does lie in such an area, there must be evidence of growth on successive imaging studies, including tumor hypervascularity, in order for such a lesion to be considered a target lesion
* The participant has a Cancer of the Liver Italian Programme (CLIP) score of 0-3
* The participant has a Child-Pugh Classification score of A or B (liver dysfunction)
* The participant has provided signed informed consent

Exclusion Criteria:

* The participant has received prior systemic chemotherapy, biologic or anti-angiogenic therapy, or investigational systemic therapy for HCC
* The participant has had bleeding from esophageal or gastric varices during the 3 months prior to study participation. Note: If the participant has any history of known esophageal varices, or evidence of esophageal varices on CT/MRI, the participant must undergo endoscopic evaluation prior to study entry (minimally invasive capsule esophageal endoscopy is an acceptable initial modality). The participant with endoscopically detected esophageal varices is eligible provided he/she meets all other entry criteria. The participant with any history or current evidence of esophageal varices must receive oral beta-blocker therapy throughout participation while on study, he/she may receive optimal endoscopic therapy as determined by the consulting gastroenterologist or hepatologist, and must undergo regular endoscopic follow-up throughout participation while on study
* The participant has acute hepatitis
* The participant has central nervous system (CNS) metastases or carcinomatous meningitis
* The participant has poorly-controlled hypertension [in other words (ie), blood pressure in abnormal range despite medical management]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Metairie, Louisiana
  - ImClone Investigational Site, Boston, Massachusetts
  - ImClone Investigational Site, Burlington, Massachusetts
  - ImClone Investigational Site, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Ramucirumab (IMC-1121B): Ramucirumab (IMC-1121B): 8 milligrams per kilogram (mg/kg) administered intravenously over 1 hour, every 2 weeks. Treatment continued until there was evidence of disease progression, intolerable toxicity, or other withdrawal criteria were met.
Period: Overall Study
Arm/Group | Ramucirumab (IMC-1121B)
Started | 42
Received at Least 1 Dose of Study Drug | 42
Completed | 40
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of ramucirumab.
Arm/Group | Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 42
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 27 (10.70)
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  Race Other: Hispanic | 1
  Race Other: Black and Asian | 1
  Race Other: Greek | 1
Region of Enrollment [Number; unit: participants]
  United States | 42
Child-Pugh Score [Number; unit: participants] — The Child-Pugh classification was used to assess the prognosis of chronic liver disease. The score employed 5 clinical measures of liver disease: encephalopathy, ascites, albumin, prothrombin time, and bilirubin. Each measure was scored from 1 (normal) and 3 (most severe derangement). The total score for the Child-Pugh assessment was calculated as the sum of the 5 contributing scores with a total possible score of 15. Chronic liver disease was classified into Child-Pugh classes A to C, employing the total score from above: 5-6=Class A; 7-9=Class B; 10-15=Class C.
  participants
    A | 31
    B | 11
Barcelona Stage [Number; unit: participants] — Barcelona Clinic Liver Cancer stage A, B, C [Franca AV et al., Braz J Med Biol Res. 2004;37(11):1689-1705]. Based on tumor burden (TB, amount of cancer in body), Child-Pugh (CP) class, Eastern Cooperative Oncology Group performance status test (PST) functional impairment [0 (Fully Active) to 5 (Death)]. Stage A [TB=single nodule or 3 nodules <3 cm, CP=A or B, PST=0 (fully active)]. Stage B (TB=single nodule >5 cm or multinodular, CP=A or B, PST=0). Stage C [TB=vascular invasion and/or metastasis, CP=A or B, PST=1 or 2 (ambulatory, restricted work activity or ambulatory, no work activity)].
  participants
    A | 2
    B | 4
    C | 36
Macrovascular Invasion [Number; unit: participants] — The number of participants with macrovascular invasion (gross vascular invasion of major portal or hepatic veins) present, absent, not available, or missing.
  participants
    Present | 7
    Absent | 32
    Not Available | 2
    Missing | 1
Extrahepatic Metastasis Status [Number; unit: participants] — The number of participants with extrahepatic metastasis (metastases originating or occurring outside the liver) present or absent.
  participants
    Present | 32
    Absent | 10
Hepatitis B and C Status [Number; unit: participants] — Number of participants with hepatitis status data (N=39). Participants whose hepatitis status is hepatitis B and C positive are not counted in the hepatitis B positive or hepatitis C positive category.
  participants
    Hepatitis B Positive | 3
    Hepatitis C Positive | 19
    Hepatitis B and C Positive | 2
    Hepatitis B and C Negative | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) in Participants With Unresectable Hepatocellular Cancer Treated With the Monoclonal Antibody Ramucirumab
Description: PFS was defined as the time from the first day of therapy to the first evidence of disease progression or death from any cause. As classified according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria, disease progression was having at least a 20% increase in the sum of the longest diameter of target lesions and/or unequivocal progression of a non-target lesion and/or detection of a new lesion. Participants who were alive and without disease progression and participants who did not progress and were subsequently lost to follow-up were censored at the last objective tumor assessment.
Time Frame: First dose to date of progressive disease or death due to any cause [every 3 cycles up to 18 months (1 cycle=2 weeks)]
Population: Intent-to-treat population: Participants who received at least 1 dose of ramucirumab. The number of participants censored was 13.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 42
months | 4.0 [2.6 to 5.7]

2. Secondary Outcome: Time to Progression
Description: The time from first day of therapy to the first date of objective evidence of progressive disease (PD) by Response Evaluation Criteria In Solid Tumors (RECIST) criteria. PD was defined as having at least a 20% increase in sum of longest diameter of target lesions and/or unequivocal progression of a non-target lesion and/or detection of new lesion. Time to PD was censored at the date of death or study discontinuation.
Time Frame: First dose to date of PD [every 3 cycles up to 18 months (1 cycle=2 weeks)]
Population: Intent-to-treat population: Participants who received at least 1 dose of ramucirumab. The number of participants censored was 20.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 42
months | 4.2 [2.8 to 8.4]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was the duration from first dose to death due to any cause. OS was censored at last contact date for participants who were alive at the end of follow-up period or lost to follow-up.
Time Frame: First dose to death due to any cause up to 37.5 months
Population: Intent-to-treat population: Participants who received at least 1 dose of ramucirumab. The number of participants censored was 10.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 42
months | 12.0 [6.1 to 19.7]

4. Secondary Outcome: Percentage of Participants With Complete Response or Partial Response (Objective Response Rate)
Description: Objective response rate (ORR) was defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR). As classified according to Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria, CR was the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm) and normalization of tumor marker level of non-target lesions. PR was having at least a 30% decrease in sum of longest diameter of target lesions.
Time Frame: First dose to date of objective progressive disease (PD) or death up to 18 months
Population: Intent-to-treat population: Participants who received at least 1 dose of ramucirumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 42
percentage of participants | 9.5 [2.7 to 22.6]

5. Secondary Outcome: Duration of Response
Description: Duration of response was the interval from the date of initial documented response [complete response (CR) or partial response (PR)] to the first documented date of disease progression, initiation of other (or additional) antitumor therapy was first reported, or death due to any cause. As classified according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria, CR was the disappearance of all target lesions, PR was having at least a 30% decrease in the sum of the longest diameter of target lesions, and disease progression was having at least a 20% increase in the sum of the longest diameter of target lesions and/or unequivocal progression of a non-target lesion and/or detection of a new lesion. Data were censored for participants who did not progress or die.
Time Frame: Time of first response (CR or PR) to disease progression, or death due to any cause [every 3 cycles up to 18 months (1 cycle=2 weeks)]
Population: Participants who received at least 1 dose of ramucirumab and had a CR or PR. The number of participants censored 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 4
months | 14.1 [4.3 to 14.1]

6. Secondary Outcome: Number of Participants With Serum Anti-Ramucirumab Antibodies
Time Frame: Prior to dosing at baseline, Cycles 4 and 7, and 30 days after end of therapy (1 cycle=2 weeks)
Population: Intent-to-treat population: Participants who received at least 1 dose of ramucirumab.
Measure: Number; unit: participants
Arm/Group | Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 42
participants | 6

7. Secondary Outcome: Number of Participants With Drug-Related Treatment-Emergent Adverse Events
Description: Data presented are the number of participants who experienced treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), Grade 3 or higher TEAEs, or adverse events (AEs) leading to discontinuation of treatment that were considered by the investigator to be related to ramucirumab. A summary of SAEs and other nonserious AEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: First dose to 37.5 months
Population: Intent-to-treat population: Participants who received at least 1 dose of ramucirumab.
Measure: Number; unit: participants
Arm/Group | Ramucirumab (IMC-1121B)
Number analyzed (Participants) | 42
participants
  Related TEAE | 41
  Related SAE | 9
  Related Grade 3 or higher TEAE | 14
  Related AE leading to discontinuation | 6

ADVERSE EVENTS:
Arm/Group | Ramucirumab (IMC-1121B)
Serious Adverse Events (participants affected / at risk) | 24/42
Other Adverse Events (participants affected / at risk) | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (IMC-1121B) (N=42)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) — Event resulted in 1 death
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
CHILLS (General disorders) | 1 (1)
DISEASE PROGRESSION (General disorders) | 1 (1) — Event resulted in death
FATIGUE (General disorders) | 2 (2)
INFUSION RELATED REACTION (General disorders) | 2 (2)
PYREXIA (General disorders) | 2 (2)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) — Event resulted in death
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Event resulted in death
ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 (2) — Event resulted in death
SYNCOPE (Nervous system disorders) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOSPITALISATION (Surgical and medical procedures) | 1 (1)
LIVER TRANSPLANT (Surgical and medical procedures) | 1 (1)
ARTERIOSCLEROSIS (Vascular disorders) | 1 (1) — Event resulted in death
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 3 (3)
HYPOTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (IMC-1121B) (N=42)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3 (3)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 8 (9)
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 (8)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 (8)
ASCITES (Gastrointestinal disorders) | 5 (9)
CONSTIPATION (Gastrointestinal disorders) | 7 (11)
DIARRHOEA (Gastrointestinal disorders) | 14 (22)
DYSPEPSIA (Gastrointestinal disorders) | 3 (3)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 15 (18)
VOMITING (Gastrointestinal disorders) | 5 (5)
ASTHENIA (General disorders) | 3 (3)
CHILLS (General disorders) | 3 (4)
FATIGUE (General disorders) | 28 (37)
INFUSION RELATED REACTION (General disorders) | 5 (7)
OEDEMA PERIPHERAL (General disorders) | 14 (19)
PYREXIA (General disorders) | 3 (3)
WEIGHT DECREASED (Investigations) | 8 (11)
ANOREXIA (Metabolism and nutrition disorders) | 11 (11)
DEHYDRATION (Metabolism and nutrition disorders) | 5 (7)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 4 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (6)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4)
DIZZINESS (Nervous system disorders) | 5 (5)
HEADACHE (Nervous system disorders) | 16 (19)
HYPOAESTHESIA (Nervous system disorders) | 3 (4)
ANXIETY (Psychiatric disorders) | 7 (8)
INSOMNIA (Psychiatric disorders) | 7 (7)
RENAL FAILURE (Renal and urinary disorders) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 (9)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 6 (8)
HYPERTENSION (Vascular disorders) | 16 (18)
HYPOTENSION (Vascular disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The duration of response results should be interpreted with caution since the sample size for this analysis was very small (2 participants).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.